CLINICAL TRIAL: NCT03761914
Title: A Phase 1/2 Study of Galinpepimut-S in Combination With Pembrolizumab (MK 3475) in Patients With Selected Advanced Cancers
Brief Title: Galinpepimut-S in Combination With Pembrolizumab in Patients With Selected Advanced Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sellas Life Sciences Group (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); LumaBridge (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLS17-201/MK3475-770
Record Dates: First submitted 2018-11-28; First posted 2018-12-03 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Acute Myelogenous Leukemia; Ovarian Cancer; Colorectal Cancer; Triple-negative Breast Cancer; Small-cell Lung Cancer
Keywords: peptide vaccine; immuno-oncology; WT1-expressing tumors; galinpepimut-S; pembrolizumab; PD1 inhibitor; checkpoint inhibitor; combination immunotherapy; heteroclitic; multivalent; off-the-shelf vaccine; HLA allele; WT1 vaccine; SLS-001; WT1 analog peptide vaccine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Ovarian Neoplasms; Colorectal Neoplasms; Triple Negative Breast Neoplasms; Small Cell Lung Carcinoma | interventions — pembrolizumab; Monatide (IMS 3015); Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Intervention Model Description: Phase 1/2, open-label, non-comparative, multicenter, multi-arm study (basket-type)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Colorectal Cancer (CRC) - opened but since only one subject enrolled, not included for analyses (Experimental): * N=20 (planned);
  * Metastatic CRC previously treated with ≥ 2 lines of prior systematic chemotherapies
  * Galinpepimut-S + Montanide + GM-CSF + pembrolizumab
  Interventions: Biological: galinpepimut-S; Biological: pembrolizumab; Other: Montanide; Biological: GM-CSF
- Ovarian Cancer (OvC) (Experimental): * N=20 (planned);
  * Metastatic platinum-resistant or refractory OvC previously treated with ≥1 line of prior platinum-containing therapy
  * Galinpepimut-S + Montanide + GM-CSF + pembrolizumab
  Interventions: Biological: galinpepimut-S; Biological: pembrolizumab; Other: Montanide; Biological: GM-CSF
- Small Cell Lung Cancer (SCLC) - not opened (Experimental): * N=20 (planned);
  * Advanced SCLC previously treated with one line of prior systemic chemotherapy
  * Galinpepimut-S + Montanide + GM-CSF + pembrolizumab
  Interventions: Biological: galinpepimut-S; Biological: pembrolizumab; Other: Montanide; Biological: GM-CSF
- Triple Negative Breast Cancer (TNBC) - not opened (Experimental): * N=15 (planned);
  * TNBC previously treated with one line of prior systemic chemotherapy
  * Galinpepimut-S + Montanide + GM-CSF + pembrolizumab
  Interventions: Biological: galinpepimut-S; Biological: pembrolizumab; Other: Montanide; Biological: GM-CSF
- Acute Myelogenous Leukemia (AML) - not opened (Experimental): * N=15 (planned);
  * AML (any age) who are not eligible for allogeneic hematopoietic stem cell transplant and have been able to achieve partial response (PR) while receiving frontline therapy with hypomethylating agents (HMAs)
  * Galinpepimut-S + Montanide + GM-CSF + pembrolizumab
  Interventions: Biological: galinpepimut-S; Biological: pembrolizumab; Other: Montanide; Biological: GM-CSF

INTERVENTIONS:
Biological: galinpepimut-S — * Induction phase: the first two GPS + Montanide injections are administered Q3W on Week 0 and Week 3. Thereafter, GPS + Montanide is co-administered with pembrolizumab Q3W (Weeks 6, 9, 12, 15, 18).
  * Early immune booster phase: A single administration of pembrolizumab (Week 21), and then GPS + Montanide resumes Q3W for six additional doses (Weeks 24, 27, 30, 33, 36, 39).
  * Following the early immune booster, there is a 12-week interval of pembrolizumab administration (Weeks 42, 45, 48, 51), and then GPS is resumed every 12 weeks for an additional four doses.
  * After 84 weeks, participants who had not progressed will continue in the study and be treated with pembrolizumab alone.
  Other Names: SLS-001; GPS; WT1 Analog Peptide Vaccine
Biological: pembrolizumab — Pembrolizumab is administered at a dose of 200 mg intravenously every 3 weeks on Day 1 of each cycle (3-week cycles) starting on Study Week 6 and continuing for up to 2 years thereafter (Study Week 108). Pembrolizumab is to be administered no earlier than 30 minutes after the administration of GPS on Day 1 of each cycle.
  Other Names: MK-3475; Keytruda
Other: Montanide — Adjuvant
Biological: GM-CSF — Participants receive 70 μg GM-CSF SC on Day -2 and on Day 1 before each GPS injection. The GM-CSF injections occur at the same anatomical site of the next planned study treatment injection.
  Other Names: sargramostim

SUMMARY:
To evaluate the safety, tolerability, and anti-tumor activity of galinpepimut-S in combination with pembrolizumab in patients with selected advanced cancers.

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, non-comparative, multicenter, multi-arm (basket-type) study of galinpepimut-S (a multivalent WT1 analog peptide vaccine) in combination with the programmed death-1 (PD1) inhibitor pembrolizumab, in patients with metastatic colorectal cancer (mCRC), metastatic ovarian cancer (mOvC), advanced small-cell lung cancer (SCLC), triple-negative breast cancer (TNBC), and acute myeloid leukemia (AML).

Additional details of tumors and prior therapies: mCRC treated with at least two prior lines, mOvC treated with at least one prior line, SCLC treated with one prior line, TNBC treated with at least one prior line, and AML unable to attain a morphological partial response after hypomethylating agents and who are not eligible for allogeneic hematopoietic stem cell transplant.

The primary objectives of the study are to assess the safety, tolerability, and anti-tumor activity of galinpepimut-S in combination with pembrolizumab. The secondary and exploratory objectives include duration of response, overall survival, and progression-free survival.

The study will enroll approximately 90 patients at up to 20 centers in the United States.

The first two galinpepimut-S injections will initially be administered as monotherapy every three weeks (Week 0 and Week 3). Thereafter, galinpepimut-S will be co-administered with pembrolizumab every three weeks for four additional administrations (for the galinpepimut-S initial immunization induction phase series; weeks 6-15) to coincide with the per label pembrolizumab dosing frequency. After that, there will be one un-paired administration of pembrolizumab (week 18), and then galinpepimut-S will be resumed Q3W for six additional doses (early immune booster phase; weeks 21-36).

At the end of this phase, there will be a 12-week interval where three unpaired administrations of pembrolizumab will occur (weeks 39-45), and then galinpepimut-S will be resumed on an every 12-week schedule for four additional doses (late immune booster phase; weeks 48-84). After 84 weeks, continuing non-progressed patients will be treated with pembrolizumab alone up until week 111.

Pembrolizumab will be administered at a dose of 200 mg intravenously Q3W on Day 1 of each cycle (three week cycles) starting on Study Week 6 and continuing for up to two years thereafter (Study Week 111). Galinpepimut-S will be administered 30-60 minutes after the completion of IV infusion of pembrolizumab on Day 1 of each cycle during which the two drugs are being co-administered.

ELIGIBILITY:
Inclusion Criteria:

* Is willing and able to understand and provide signed informed consent for the study that fulfills IRB guidelines
* Male or female patients >18 years of age on the day of signing informed consent
* Histologically or cytologically-confirmed advanced or metastatic solid tumors who have disease progression after treatment with available therapies for metastatic disease that are known to confer clinical benefit, or are intolerant to treatment, or refuse standard treatment in the context of the particular line of treatment or, specifically for AML, demonstrate as their best response after 4 cycles of HMA therapy the status of "partial response" per European LeukemiaNet (ELN) criteria and meet the additional specified requirements for the cohort of the study they will enroll into.
* All patients in the solid tumor arms will be tested for WT1 expression via IHC in their initial primary tumor OR recent biopsy of metastatic disease at the time of screening for study entry. Specifically for AML, patients will be tested for WT1 expression via IHC in their leukemic blasts either in the BM or PB. Assessment of WT1 expression positivity will be performed via central review prior to study entry.
* Patients may have received a specific maximum allowable number of prior lines of therapy for metastatic disease, as follows: CRC: 2 or 3 lines; OvC: 1 or 2 lines; SCLC: 1 line; TNBC: 1 line; and AML: 1 line (allo-SCT-eligible status not allowed)
* For solid tumor arms: patients must measurable disease based on RECIST v1.1 as determined by the local study team.
* For AML arm, eligibility is defined as:

  1. Prior frontline (1st line) with HMAs since initial AML diagnosis;
  2. Prior cytoreductive therapy with hydroxyurea or leukapheresis at the time of initial diagnosis, with subsequent immediate seamless transitioning to HMA therapy
  3. History of induction early failure after initial therapy with up to 2 cycles of standard chemotherapy ("7+3" or similar regimen), with subsequent immediate seamless transitioning to HMA therapy as long as patients have achieved PR as their best observable response after 4 cycles of HMA therapy; HMA therapy continues throughout the trial period.
* Resolution of toxicity effect(s) from most recent prior chemotherapy to Grade 1 or less (except alopecia). If the patient received major surgery or radiation therapy of > 30 Gy, they must have recovered from the toxicity and/or complications from the intervention.
* (ECOG) performance status of 0 or 1.
* For women of child-bearing potential, agreement to use adequate birth control (abstinence, hysterectomy, bilateral oophorectomy, bilateral tubal ligation, oral contraception, IUD, or use of condoms or diaphragms)
* Male patients of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 4 months following the last study treatment.
* Have adequate organ function as defined:

  * Absolute neutrophil count (ANC) ≥1500/µL
  * Platelets ≥100,000/µL
  * Hemoglobin (Hb) ≥9.0 g/dL or ≥5.6 mmol/L (N.B.: Hb criterion must be met without erythropoietin dependency and without packed red blood cell transfusion within last 2 weeks)
  * Creatinine ≤1.5 × upper limit of normal (ULN) OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥30 mL/min for subjects with creatinine levels >1.5 × institutional ULN
  * Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for subjects with total bilirubin levels >1.5 × ULN
  * AST (SGOT) and ALT (SGPT) ≤2.5 × ULN OR ≤5 × ULN for subjects with liver metastases
  * International normalized ratio (INR) OR prothrombin time (PT) and Activated partial thromboplastin time (aPTT) ≤1.5 × ULN, unless subjects are receiving anticoagulant therapy as long as PT or aPTT is within the therapeutic range of intended use of anticoagulants

Additional Inclusion Criteria for Selected Tumor Types:

(i).Colorectal Cancer (third/fourth line)

* Histologically or cytologically documented adenocarcinoma of colon or rectum at the time of initial presentation.
* Metastatic CRC with documented disease progression (per standard criteria) after the last administration of standard therapies or intolerance to standard therapies (and approved therapies must have included all the following a fluoropyrimidine, oxaliplatin, irinotecan, bevacizumab, and, if KRAS wild-type, cetuximab or panitumumab). Prior use of and failure after regorafenib or trifluridine/tipiracil is allowed but not mandated.

(ii). OvC (second/third line)

* Histologically diagnosed ovarian, fallopian tube or primary peritoneal cancer at the time of initial presentation.
* Patients will have either relapsed or be disease resistant to their prior therapy. Interval surgery is permitted, but patients must have objective evidence of disease on computed tomography (CT)or magnetic resonance imaging (MRI), with concomitant CA-125 increase and/or biopsy showing OvC (only for recurrent disease).
* Patients should have received platinum-containing chemotherapy and been designated as harboring platinum-refractory or -resistant disease. Additionally, all eligible subjects should have either received (or been offered) bevacizumab therapy, and those with BRCA germline mutations (gBRCA mut) should have been offered therapy with poly-ADP ribose polymerase (PARP) inhibitors (olaparib, rucaparib or niraparib).

(iii). SCLC (second line)

* Histologically or cytologically confirmed SCLC based on biopsy of the tumor at initial presentation.
* Asymptomatic or treated brain metastases are allowed.
* Patients must have measurable disease (by CT or MRI) after they progressed or were resistant to 1 prior systemic therapy.

(iv). TNBC (second line)

* Histologically proven metastatic breast carcinoma with triple negative receptor status.
* TNBC status is defined as estrogen and progesterone receptor negative by IHC, and human epidermal growth factor receptor 2 [HER2] negative by IHC AND HER2 gene non-amplified by fluorescence in situ hybridization [FISH], per standard criteria. Patients who are weakly positive for the estrogen or progesterone receptor (i.e., < 5%) are eligible.
* Patients must have measurable disease(by CT or MRI) after they progressed or were resistant to 1 prior systemic therapy.
* Patients have undergone second-line therapy after residual or recurrent disease after first-line therapy. The latter may have included:

  1. Neoadjuvant therapy if macroscopic disease was still present after surgery OR
  2. Adjuvant therapy, but only if the macroscopic relapse occurred > 6 months from the start of study treatment with pembrolizumab.

  (v). AML
* Pathologically or morphologically confirmed de novo or secondary AML at the time of initial diagnosis.
* Achievement of no better than morphologic PR, as defined initially by the AML Working Group criteria (Cheson et al,2003), and also quoted in the more recent ELN criteria (Döhner et al, 2010),while on active treatment with HMAs.
* AML patients are eligible only if they received first-line therapy with HMAs (decitabine or azacytidine) for 4 cycles and achieved only PR at the end of cycle 4.
* AML patients must remain on HMA therapy throughout the trial.

Exclusion Criteria:

* Presence of disease that is suitable for local or regional therapy administered with curative intent.
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to treatment.

  * N.B.: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.
  * N.B.: If the subject underwent major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
* Has received prior radiotherapy within 2 weeks of the start of study treatment. Subjects must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137) and was discontinued from that treatment due to a Grade 3 or higher immune-related adverse event (irAE).
* Subject currently participates in a clinical trial with another investigational agent and is receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first study treatment.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
* Has undergone prior allogeneic hematopoietic stem cell transplantation.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor. Steroids taken as short-term therapy (≤ 7 days) for antiemesis are permissible.
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years, even if currently inactive or unapparent.

  - N.B.: Specifically, AML patients with prior history of myelodysplastic syndromes or myeloproliferative neoplasms are not excluded. Participants in any of the study arms (solid tumors or AML) with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy, as well as patients with prostate cancer managed clinically with "watchful waiting" are eligible.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has known hypersensitivity to Montanide or vaccine adjuvants.
* Had a previous clinically significant systemic allergic reaction to Montanide, sargramostim (GM-CSF), or filgrastim (G-CSF).
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease-modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Subjects with known human immunodeficiency virus (HIV) and/or history of Hepatitis B or C infections, or known to be positive for Hepatitis B antigen (HBsAg)/ Hepatitis B virus (HBV) DNA or Hepatitis C Antibody or RNA are excluded. Active Hepatitis C is defined by a known positive Hep C Ab result and known quantitative HCV RNA results greater than the lower limits of detection of the assay.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator. This includes any serious, intercurrent, chronic, or acute illness, such as cardiac disease (New York Heart Association [NYHA] class III or IV), hepatic disease, or other illness considered by the investigator as an unwarranted high risk for investigational drug treatment.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
* For female subjects: Subject is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 30 days after the last dose of study treatment.
* Has had an allogeneic tissue/solid organ transplant.
* Has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (excluding GM-CSF, but including G-CSF or recombinant erythropoietin) within 4 weeks prior to first study treatment.

Additional Exclusion Criteria for Selected Tumor Types:

(i). CRC: None (ii). OvC: None (iii). SCLC: Mixed SCLC (iv). TNBC: None (v). AML:

1. Planned/anticipated HSCT (autologous or allogeneic, with any degree of match donor); acute promyelocytic leukemia (APL; M3 or any morphologic and molecular variants, inclusive); history or current diagnosis of CNS leukemia
2. Relapsed (Second line) patients

   * N.B.: Patients who received any chemotherapy ("3 + 7" or similar chemotherapy regimen) for up to 2 cycles during initial induction therapy in the first-line setting and subsequently immediately seamlessly switched to HMAs are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Sarlis, MD, PhD, Study Director — SELLAS Life Sciences Group, Inc.
Locations (12):
- United States (12):
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - Innovative Clinical Research Institute (ICRI), Whittier, California
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center, Commack, New York
  - Memorial Sloan Kettering Cancer Center, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, Nassau, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ovarian Cancer (OvC): * Metastatic platinum-resistant or refractory OvC previously treated with ≥1 line of prior platinum-containing therapy
  * Galinpepimut-S + Montanide + GM-CSF + pembrolizumab
- Colorectal Cancer (CRC): * Metastatic CRC previously treated with ≥ 2 lines of prior systematic chemotherapies
  * Galinpepimut-S + Montanide + GM-CSF + pembrolizumab
- Small Cell Lung Cancer (SCLC): * Advanced SCLC previously treated with one line of prior systemic chemotherapy
  * Galinpepimut-S + Montanide + GM-CSF + pembrolizumab
- Triple Negative Breast Cancer (TNBC): * TNBC previously treated with one line of prior systemic chemotherapy
  * Galinpepimut-S + Montanide + GM-CSF + pembrolizumab
- Acute Myelogenous Leukemia (AML): * AML (any age) who are not eligible for allogeneic hematopoietic stem cell transplant and have been able to achieve partial response (PR) while receiving frontline therapy with hypomethylating agents (HMAs)
  * Galinpepimut-S + Montanide + GM-CSF + pembrolizumab
Period: Overall Study
Arm/Group | Ovarian Cancer (OvC) | Colorectal Cancer (CRC) | Small Cell Lung Cancer (SCLC) | Triple Negative Breast Cancer (TNBC) | Acute Myelogenous Leukemia (AML)
Started | 25 | 1 (This arm only enrolled 1 subject before it was closed. Subject was not included in the efficacy or safety analyses.) | 0 (This arm was not opened) | 0 (This arm was not opened) | 0 (This arm was not opened)
Completed | 25 | 1 (This arm only enrolled 1 subject before it was closed. Subject was not included in the efficacy or safety analyses.) | 0 (This arm was not opened) | 0 (This arm was not opened) | 0 (This arm was not opened)
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only the Ovarian Cancer (OvC) arm enrolled fully. One subject enrolled in the Colorectal Cancer (CRC) arm but discontinued before efficacy could be assessed. For this reason, this subject was not included in the evaluation for efficacy or safety. The other cohorts did not open.
Groups:
- Colorectal (CRC): Metastatic CRC previously treated with ≥ 2 lines of prior systematic chemotherapies Galinpepimut-S + Montanide + GM-CSF + pembrolizumab
- Total: Total of all reporting groups
Arm/Group | Ovarian Cancer (OvC) | Colorectal (CRC) | Total
Number analyzed (Participants) | 25 | 1 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only the Ovarian Cancer (OvC) arm enrolled fully. One subject enrolled in the Colorectal Cancer (CRC) arm but discontinued before efficacy could be assessed. For this reason, this subject was not included in the evaluation for efficacy or safety. The other cohorts did not open.
  years | 63.8 (7.9) | 40 (0) | 63.8 (7.9)
Age, Continuous [Median (Full Range); unit: years] — Population: Only the Ovarian Cancer (OvC) arm enrolled fully. One subject enrolled in the Colorectal Cancer (CRC) arm but discontinued before efficacy could be assessed. For this reason, this subject was not included in the evaluation for efficacy or safety. The other cohorts did not open.
  years | 65 [50 to 76] | 40 [40 to 40] | 65 [50 to 76]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only the Ovarian Cancer (OvC) arm enrolled fully. One subject enrolled in the Colorectal Cancer (CRC) arm but discontinued before efficacy could be assessed. For this reason, this subject was not included in the evaluation for efficacy or safety. The other cohorts did not open.
  Participants
    Female | 25 | 1 | 26
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only the Ovarian Cancer (OvC) arm enrolled fully. One subject enrolled in the Colorectal Cancer (CRC) arm but discontinued before efficacy could be assessed. For this reason, this subject was not included in the evaluation for efficacy or safety. The other cohorts did not open.
  Participants
    Hispanic or Latino | 8 | 0 | 8
    Not Hispanic or Latino | 14 | 1 | 15
    Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only the Ovarian Cancer (OvC) arm enrolled fully. One subject enrolled in the Colorectal Cancer (CRC) arm but discontinued before efficacy could be assessed. For this reason, this subject was not included in the evaluation for efficacy or safety. The other cohorts did not open.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 1 | 2
    White | 19 | 0 | 19
    More than one race | 5 | 0 | 5
    Unknown or Not Reported | 0 | 0 | 0
Weight [Median (Full Range); unit: kg] — Population: Only the Ovarian Cancer (OvC) arm enrolled fully. One subject enrolled in the Colorectal Cancer (CRC) arm but discontinued before efficacy could be assessed. For this reason, this subject was not included in the evaluation for efficacy or safety. The other cohorts did not open.
  kg | 61.7 [48 to 94] | 69.5 [69.5 to 69.5] | 61.7 [48 to 94]
Height [Median (Full Range); unit: cm] — Population: Only the Ovarian Cancer (OvC) arm enrolled fully. One subject enrolled in the Colorectal Cancer (CRC) arm but discontinued before efficacy could be assessed. For this reason, this subject was not included in the evaluation for efficacy or safety. The other cohorts did not open.
  cm | 160 [150 to 172] | 169 [169 to 169] | 160 [150 to 172]
BMI [Median (Full Range); unit: kg/m^2] — Population: Only the Ovarian Cancer (OvC) arm enrolled fully. One subject enrolled in the Colorectal Cancer (CRC) arm but discontinued before efficacy could be assessed. For this reason, this subject was not included in the evaluation for efficacy or safety. The other cohorts did not open.
  kg/m^2 | 25.03 [18.6 to 34.2] | 24.3 [24.3 to 24.3] | 25.03 [18.6 to 34.2]
Baseline ECOG [Count of Participants; unit: Participants] — ECOG measures patient's functional status. Grade 0 is best, grade 5 worst. Grade 0: Fully active, able to carry on all pre-disease performance without restriction Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature Grade 2: Ambulatory and capable of all self-care but unable to carry out any work activities Grade 3: Capable of only limited self-care; confined to bed or chair more than 50% of waking hours Grade 4: Completely disabled; cannot carry on any self-care; totally confined to bed or chair Grade 5: Dead Population: Only the Ovarian Cancer (OvC) arm enrolled fully. One subject enrolled in the Colorectal Cancer (CRC) arm but discontinued before efficacy could be assessed. For this reason, this subject was not included in the evaluation for efficacy or safety. The other cohorts did not open.
  Participants
    0 | 8 | 0 | 8
    1 | 17 | 1 | 18
Lines of prior therapy [Count of Participants; unit: Participants] — The number of anti-cancer therapies that patient received before joining the study. Population: Only the Ovarian Cancer (OvC) arm enrolled fully. One subject enrolled in the Colorectal Cancer (CRC) arm but discontinued before efficacy could be assessed. For this reason, this subject was not included in the evaluation for efficacy or safety. The other cohorts did not open.
  Participants
    1 | 2 | 0 | 2
    2 | 13 | 0 | 13
    3 | 3 | 0 | 3
    4 | 1 | 1 | 2
    5 | 1 | 0 | 1
    Unknown / Not reported | 5 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) - Best Overall Response
Description: Percentage of patients who have received at least one dose of pembrolizumab and have responded (and have completed imaging requirements). Best overall response is defined as the best overall visit response in the following order: CR, PR, SD, PD, or UE as measured by RECIST 1.1
Time Frame: 33 months
Population: Participants who have received at least one dose of pembrolizumab (mITT population). Patients only enrolled in the Ovarian Cancer (OvC) arm. One subject enrolled in the Colorectal Cancer (CRC) arm but discontinued before efficacy can be assessed. The other arms/groups were removed from this study.
Measure: Count of Participants; unit: Participants
Groups:
- Colorectal Cancer (CRC): One subject enrolled but discontinued before efficacy can be assessed. For this reason, this subject was not included in the evaluation for efficacy or safety.
Arm/Group | Ovarian Cancer (OvC) | Colorectal Cancer (CRC)
Number analyzed (Participants) | 16 | 0
Participants
  Complete response | 0 | 0
  Partial response | 1 | 0
  Stable disease | 7 | 0
  Progressive disease | 8 | 0

2. Primary Outcome: Overall Response Rate (ORR) - Overall Response Rate
Description: Percentage of patients who have received at least one dose of pembrolizumab and have responded (and have completed imaging requirement). Overall response rate is defined as the proportion of participants with a best overall response of CR or PR as defined by RECIST 1.1
Time Frame: 33 months
Population: Participants who have received at least one dose of pembrolizumab (mITT population).
  Patients only enrolled in the Ovarian Cancer (OvC) arm. One subject from the Colorectal Cancer (CRC) arm enrolled but discontinued before efficacy can be assessed. The other arms/groups were removed from this study.
Measure: Count of Participants; unit: Participants
Groups:
- Colorectal Cancer: One subject enrolled but discontinued before efficacy can be assessed. For this reason, this subject was not included in the evaluation for efficacy or safety.
Arm/Group | Ovarian Cancer (OvC) | Colorectal Cancer
Number analyzed (Participants) | 16 | 0
Participants | 1 | 0

3. Other Pre Specified Outcome: Progression-free Survival (PFS) - Kaplan Meier Estimate
Description: Time from enrollment to date of first confirmed disease progression or death whichever occurred earlier
Time Frame: 33 months
Population: Participants who received at least one dose of pembrolizumab (galinpepimut-S + pembrolizumab); mITT population. Patients only enrolled in the Ovarian Cancer (OvC) arm. One subject from the Colorectal Cancer (CRC) arm enrolled but discontinued before efficacy can be assessed. The other arms/groups were removed from this study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ovarian Cancer (OvC) | Colorectal Cancer
Number analyzed (Participants) | 16 | 0
months | 2.9 [2.0 to 5.6] |

4. Other Pre Specified Outcome: Overall Survival (OS) - Kaplan Meier Estimate
Description: Time from enrollment to date of death from any cause
Time Frame: 33 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ovarian Cancer (OvC) | Colorectal Cancer
Number analyzed (Participants) | 16 | 0
months | 18.4 [8.4 to NA] — Upper 95%CI not reached due to end of study monitoring duration |

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 29 months.
Description: All patients enrolled in the Ovarian Cancer (OvC) arm except for one subject enrolled in the Colorectal (CRC) arm. The CRC arm patient was discontinued before efficacy could be assessed. For this reason, this subject was not included in the evaluation for efficacy or safety.
Groups:
- Colorectal Cancer (CRC): Metastatic CRC previously treated with ≥ 2 lines of prior systematic chemotherapies Galinpepimut-S + Montanide + GM-CSF + pembrolizumab
Arm/Group | Ovarian Cancer (OvC) | Colorectal Cancer (CRC)
All-Cause Mortality (participants affected / at risk) | 7/25 | 0/0
Serious Adverse Events (participants affected / at risk) | 5/25 | 0/0
Other Adverse Events (participants affected / at risk) | 25/25 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ovarian Cancer (OvC) (N=25) | Colorectal Cancer (CRC) (N=0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Acute kidney injury (Renal and urinary disorders) | 1 (1) | NA
Hydronephrosis (Renal and urinary disorders) | 1 (1) | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | NA
Fatigue (General disorders) | 1 (1) | NA
Sepsis (Infections and infestations) | 1 (1) | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ovarian Cancer (OvC) (N=25) | Colorectal Cancer (CRC) (N=0)
Anemia (Blood and lymphatic system disorders) | 5 (5) | NA
Vomiting (Gastrointestinal disorders) | 9 (9) | NA
Abdominal pain (Gastrointestinal disorders) | 7 (7) | NA
Nausea (Gastrointestinal disorders) | 7 (7) | NA
Abdominal distension (Gastrointestinal disorders) | 6 (6) | NA
Diarrhea (Gastrointestinal disorders) | 6 (6) | NA
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | NA
Constipation (Gastrointestinal disorders) | 5 (5) | NA
Ascites (Gastrointestinal disorders) | 4 (4) | NA
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | NA
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | NA
Fatigue (General disorders) | 8 (8) | NA
Injection site reaction (General disorders) | 6 (6) | NA
Edema peripheral (General disorders) | 4 (4) | NA
Pain (Gastrointestinal disorders) | 4 (4) | NA
Pyrexia (General disorders) | 3 (3) | NA
Influenza like illness (General disorders) | 2 (2) | NA
Hypersensitivity (Immune system disorders) | 2 (2) | NA
Urinary tract infection (Infections and infestations) | 3 (3) | NA
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | NA
Dehydration (Metabolism and nutrition disorders) | 2 (2) | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | NA
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | NA
Headache (Nervous system disorders) | 8 (8) | NA
Aphasia (Nervous system disorders) | 5 (5) | NA
Insomnia (Psychiatric disorders) | 2 (2) | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | NA
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | NA
Hypotension (Vascular disorders) | 2 (2) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT03761914/Prot_SAP_001.pdf